CLINICAL TRIAL: NCT02168166
Title: Short-Term Executive Functioning Training
Brief Title: Short-term Working Memory and Executive Training
Acronym: STExFx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Christopher Bowie, Dr., Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GPSYC-651-14
Record Dates: First submitted 2014-06-16; First posted 2014-06-20 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Psychotic Disorders
Keywords: Neurological Disorders; Neuroscience; Neuropsychology; EEG; Cognitive remediation; Cognitive Response
MeSH Terms: conditions — Psychotic Disorders; Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Executive Function Training (Active Comparator): Two weeks of training of cognitive domain of executive functioning
  Using online program (Scientific Brain Training Pro)
  Four exercises
  Interventions: Behavioral: Executive Function Training
- Placebo Training (Placebo Comparator): Two weeks of training with exercises not affecting working memory, information processing speed, or cognitive load
  Exercises maintain other traditional progressive aspects to preserve appearance of dynamic titration of difficulty levels
  Using online program (Scientific Brain Training Pro)
  Four exercises
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Executive Function Training
  Arms: Executive Function Training
Behavioral: Placebo — Placebo version of executive function training
  Arms: Placebo Training

SUMMARY:
Cognitive remediation (CR) therapies refer to a number of recent developments to use behavioural strategies to improve neurocognitive abilities and improve everyday functioning in mental disorders such as schizophrenia, bipolar disorder, and depression. In this study, we aim to examine whether we can observe CR effects on measures of neuroplasticity, cognition, and functioning when using a rigorous control comparison group. We hypothesize that the active group will exhibit improvements in executive functioning composite scores, improved EEG theta-gamma frequency modulation, and increased EEG alpha power compared to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of a chronic mental disorder (defined herein as bipolar disorder, major depressive disorder, or a schizophrenia-spectrum disorder)
* between the ages of 18 and 65
* speak and read fluent English
* able to use a computer

Exclusion Criteria:

* active substance abuse or dependence diagnosis
* sensory or motor issues that would preclude completion of study procedures
* enrollment in a cognitive remediation program or use of cognitive training programs (e.g. lumosity.com) within the past 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-05; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline executive functioning composite score at post-treatment assessment | Pre-training assessment (Week 1) and post-training assessment (Week 4)
  Composite score based on four tests of cognition

SECONDARY OUTCOMES:
Change from baseline EEG theta-gamma frequency modulation at post-treatment assessment | Pre-training assessment (Week 1) and post-training assessment (Week 4)
  Predicted to improve in active CR (cognitive remediation) condition compared to placebo CR
Change from baseline EEG alpha power at post-treatment assessment | Pre-training assessment (Week 1) and post-training assessment (Week 4)
  Predicted to increase in active CR (cognitive remediation) condition compared to placebo CR

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Bowie, PhD, CPsych, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada